CLINICAL TRIAL: NCT03693586
Title: Study to Determine the Hepatitis C Virus Infection Prevalence Among Patients Attended Primarily for Vasculitis and Other Potential Extrahepatic Manifestations
Brief Title: Study to Determine the Hepatitis C Virus Infection Prevalence Among Patients Attended Primarily for Vasculitis
Status: Completed | Type: Observational
Sponsor: Hospital General de Mexico (Other Government)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, MARIA DE FATIMA HIGUERA DE LA TIJERA, Head of Gastroenterology and Hepatology Department, Hospital General de Mexico
Other Study IDs: DI/18/107/03/071
Record Dates: First submitted 2018-09-19; First posted 2018-10-03 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Chronic Hepatitis c; Vasculitis
Keywords: seroprevalence; viral load; chronic hepatitis c; vasculitis
MeSH Terms: conditions — Hepatitis C, Chronic; Vasculitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic hepatitis C infection (CHC) is usually asymptomatic; nevertheless, there are studies that show that up to two thirds of patients may present some type of extrahepatic manifestation. The most frequent extrahepatic manifestation is type II mixed cryoglobulinemia (MCG-II) and clinically the most common presentation is leukocytoclastic vasculitis (LCV) with palpable purpura that affects the lower extremities. It is estimated that up to 80% of MCG-II cases are due to CHC. Also, previous studies have demonstrated that CHC prevalence is higher in patients with autoimmune diseases compared with general population. Therefore, if vasculitis is an extrahepatic manifestation of CHC, then the prevalence of CHC infection in this group of patients could be higher than the prevalence reported in general population.

The aim of the study is to know the prevalence of CHC, determined by serological rapid test for hepatitis C screening, then all positive cases will be confirmed by quantitative viral load, in patients who consult primarily to a rheumatology department for "vasculitis" or other potential hepatitis C extrahepatic manifestations (rheumatological conditions).

DETAILED DESCRIPTION:
1. Introduction.

   The prevalence of Hepatitis C determined by serological test to detect antibodies against the hepatitis C virus (HCV) is around 1.4% in Mexico, being slightly higher in the north (2.0%) than in the south (1.5%). ) and the entities of the center (1.1%) of the country. However, there are high risk groups where the prevalence is much higher, for example, among intravenous drug users such as heroin, it is estimated that prevalence of hepatitis C is as high as 11.7%, with an interval ranging from 2.7 to 39.1% .

   Recently, the Global Prevalence study of HCV - Polaris Observatory at American Association for de the Study of Liver (AASLD), has documented that the prevalence in Mexico determined by viral load quantification (which is the most specific study) ranges from 0.0 to 0.6%, being higher in the North, than in the Center and in the South of the country.

   Although it is classically considered that chronic hepatitis C infection (CHC) is usually asymptomatic, there are studies that show that up to two thirds of patients may present some type of extrahepatic manifestation. The most frequent extrahepatic manifestation is type II mixed cryoglobulinemia (MCG-II) and clinically the most common presentation is leukocytoclastic vasculitis (LCV) with palpable purpura that affects the lower extremities. It is estimated that up to 80% of MCG-II cases are due to CHC. The prevalence of CHC infection has been reported in higher numbers in patients with LCV than in the general population. A multinational study in 2009, found that the prevalence of anti-HCV antibodies specifically in patients consulting for "autoimmune diseases" was as high as 8.7%, compared to healthy subjects (general population) where it was 0.4%. In this study, the diagnosis of CHC with determination of viral load or genotype was not confirmed.

   In another study, conducted in Brazil, which included 367 patients with rheumatological diseases, the prevalence of CHC, confirmed with viral load determination, was 1.9%, also higher than that reported in the open population in that country. The difference remarkable in the prevalences reported by serological tests and by viral load, particularly in patients with autoimmune diseases, can be explained because patients with autoimmune diseases have autoantibodies that can generate cross reactions and result in false positives, for this reason, in the presence of a positive result in these tests, must always be confirmed with the gold standard that is the quantification of viral load.
2. Research question.

   Will the prevalence of hepatitis C determined by quantitative viral load be higher in patients who consult as first-line for vasculitis, a possible extrahepatic manifestation of HCV, compared to that reported in the general Mexican population?
3. Approach of the problem.

   Previous studies in other countries show that the prevalence of HCV infection is higher in patients with autoimmune clinical manifestations, specifically vasculitis, since this may be extrahepatic manifestation of HCV, compared to the general population.

   In Mexico, the prevalence of HCV in the population of patients with "vasculitis" has never been evaluated.

   Since the timely detection of chronic HCV infection requires a high degree of suspicion based on the patient's risk factors, and since their symptoms are totally nonspecific, and knowing that vasculitis associated with MCG-II is the most extrahepatic manifestation common of HCV, the investigators consider relevant to perform an HCV screening in this group of patients.
4. Justification.

   At present, HCV infection is curable with high effectiveness, achieving the sustained viral response in more than 95% of cases with the new direct antiviral agents. Early diagnosis depends on the patient having access to an effective treatment and that achieving a virological cure achieves a favorable prognosis for function and life.
5. Hypothesis.

   If vasculitis is an extrahepatic manifestation of HCV, then the prevalence of chronic HCV infection in this group of patients will be higher than the prevalence reported in the general population.
6. Objectives.

   General: To know the real prevalence of hepatitis C determined by quantitative viral load in patients who consult for the first intention to a rheumatology department for "vasculitis and with a positive result in the serological HCV screening test".

   Specific(1): To describe the clinical characteristics of hepatic and extrahepatic manifestations of patients with "vasculitis" detected with Hepatitis C.

   Specific (2): To determine the real prevalence of hepatitis C determined by quantitative viral load in patients who consult for other rheumatological conditions (non-vasculitis) with a positive result in the serological HCV screening test.
7. Material and methods.

   1. Type and design of the study: Observational study, case series, descriptive and analytical.
   2. Inclusion criteria: Patients who first attend to a Rheumatology department, to be evaluated for diagnosis of "vasculitis under study" or "vasculitis of origin to be determined" or "rheumatological condition for study".
   3. Exclusion criteria: Patients who do not wish to participate in the study.
   4. Elimination criteria: Patients who do not have a complete clinical file.
   5. Population and sample size:

      Population: All patients who first attend to a Rheumatology department, to be evaluated for diagnosis of "vasculitis under study" or "vasculitis of origin to be determined" or "rheumatological condition for study".

      Sample size: Assuming a prevalence of between 5 to 10%, in this specific population, a total of 1000 patients need to be evaluated, to find between 50 to 100 patients with chronic HCV infection.
   6. Data collection and Procedures: The investigators will obtain the informed consent from patients; demographic, clinical, biochemical data of the clinical file will be collected. A quick test will be taken in the office for HCV detection, if it is negative, it is recorded in the data collection form and the patient will be discharged from this clinical study to continue the usual care in Rheumatology. If this test is positive, the patient will be given a request for viral load and genotype and an appointment will be made for follow-up of the case in the Liver Clinic.
8. Relevance and expectations

This will be the first study in Mexico to characterize a population that suffers from vasculitis, the most common extrahepatic manifestation related to MCG-II in patients with HCV, and other rheumatological conditions, as potential extrahepatic manifestations of CHC.

This study will allow to know the prevalence in this special group of patients, in addition to the research purposes that fall within this prevalence study, patients will have access to a detection and treatment program in a timely manner.

ELIGIBILITY:
Inclusion Criteria:

* patients who primarily consults to a rheumatology department for vasculitis and agree to be evaluated through a questionaire to identify risk factors for hepatitis C and who also agree to be screened with a serological rapid test for hepatitis C.

Exclusion Criteria:

* patients who decline to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who primarily consults to a rheumatology department for vasculitis and agree to be evaluated through a questionaire to identificate risk factors for hepatitis C and who also agree to be screened with a serological rapid test for hepatitis C
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
seropositive for hepatitis C | 1 year
  serological rapid test screening for hepatitis C

SECONDARY OUTCOMES:
confirmation of a hepatitis C case | 1 year
  viral load and genotypification

CONTACTS AND LOCATIONS:
Overall Officials: FATIMA HIGUERA-DE LA TIJERA, MSc., Principal Investigator — Hospital General de México
Locations (1):
- Hospital General de Mexico, Mexico City, Mexico